CLINICAL TRIAL: NCT01613534
Title: Argon Plasma Coagulation Plus Placebo or Oral Sucralfate for Chronic Radiation Proctopathy: a Randomized Placebo Controlled Trial
Brief Title: Combined Therapy in Radiation Proctopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Medical Centre for Postgraduate Education (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 501-2-1-09-14/03
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Radiation Proctitis
Keywords: chronic radiation proctopathy; argon plasma coagulation; sucralfate
MeSH Terms: interventions — Sucralfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- APC plus oral sucralfate (Experimental): Argon plasma coagulation treatment followed by oral sucralfate (6 grams b.i.d.) administration for four weeks.
  Interventions: Drug: Sucralfate
- APC plus placebo (Placebo Comparator): Argon plasma coagulation treatment followed by placebo administration for four weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sucralfate — Argon plasma coagulation treatment followed by oral sucralfate (6 grams b.i.d.) for four weeks
  Other Names: Carafate; Ulgastran
  Arms: APC plus oral sucralfate
Drug: Placebo — Argon plasma coagulation treatment followed by placebo administration for four weeks
  Arms: APC plus placebo

SUMMARY:
The aim of this study was to compare the efficacy and safety of two treatment regimens: argon plasma coagulation (APC) alone and APC in combination with sucralfate administered for chronic hemorrhagic radiation proctopathy.

DETAILED DESCRIPTION:
Chronic radiation proctopathy (CRP) or proctosigmoiditis is a late complication of pelvic radiotherapy. Symptoms, including diarrhea, rectal bleeding, urgency, and tenesmus, are difficult to treat and adversely impact patient quality of life. Various treatments directed at the reduction of blood loss and improvement of other symptoms have been evaluated, with the most encouraging results reported for two methods: endoscopic argon plasma coagulation (APC) of radiation-induced abnormal vessels in the rectal mucosa, and administration of sucralfate, a drug believed to enhance the mucosal defense and healing when administered orally or rectally. Adequately powered randomized trials comparing various treatments are lacking, and an optimal management strategy has yet to be determined. To address this issue, we conducted a single-center, randomized, placebo-controlled, double-blind study comparing the efficacy and safety of APC alone and APC in combination with sucralfate administered orally.

ELIGIBILITY:
Inclusion Criteria:

* radiotherapy due to pelvic tumors completed at least three months prior to enrollment
* presence of rectal bleeding
* radiation-induced telangiectasia in the rectum and/or sigmoid colon on endoscopy
* informed written consent to participate in the study

Exclusion Criteria:

* history of clinically significant rectal bleeding prior to radiotherapy
* conditions predisposing the patient to rectal bleeding including inflammatory bowel disease, tumors of the large bowel, intestinal vascular lesions (other than radiation-induced telangiectasia), and diversion of the fecal stream
* sucralfate treatment during the two weeks prior to enrollment
* renal insufficiency (creatinine level ≥2 mg/dl)
* concurrent chemotherapy
* concurrent therapy with tetracycline, fluoroquinolones, or antimycotic drugs (because of drug interaction)
* concurrent therapy with oral anticoagulants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2003-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
change in disease severity scores, as assessed using our three-item symptom scale | baseline vs. 16 week
  Three-item symptom scale Diarrhea - score 1: 1-3 stools/24 h; 2: 4-6 stools/24 h; 3 >6 stools/24 h Bleeding - score 0: No blood; 1: Blood on toilet paper or stool; 2: Blood in toilet bowl; 3: Heavy bleeding with clots; 4: Bleeding requiring transfusions Tenesmus/rectal pain - score 0: Absent; 1: Mild tenesmus not requiring any drug; 2: Tenesmus requiring analgesics/antispasmodics; 3: Severe tenesmus requiring everyday use of analgetics/antispasmodics.

SECONDARY OUTCOMES:
change in endoscopic severity score | baseline vs. week 8 and week 16
  Endoscopic severity score of chronic radiation proctopathy:
  Normal, score 0 - Normal mucosa Mild, score 3 - Erythema and/or teleangiectasia, edema, thickening, pallor of mucosa Moderate, score 6 - Above plus friability Severe, score 9 - Ulceration and/or necrosis
change in disease severity score | baseline vs. week 52
  disease severity score as in primary outcome measure
complication rate | baseline to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena R Chruscielewska-Kiliszek, MD, PhD, Principal Investigator — Medical Centre for Postgraduate Education
Locations (1):
- Department of Gastroenterology and Hepatology, Medical Center for Postgraduate Education and Department of Gastroenterology, Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Derived] Chruscielewska-Kiliszek MR, Regula J, Polkowski M, Rupinski M, Kraszewska E, Pachlewski J, Czaczkowska-Kurek E, Butruk E. Sucralfate or placebo following argon plasma coagulation for chronic radiation proctitis: a randomized double blind trial. Colorectal Dis. 2013 Jan;15(1):e48-55. doi: 10.1111/codi.12035. PMID 23006660